CLINICAL TRIAL: NCT01730638
Title: Pharmacokinetic and Imaging Optimization Study of Pretargeted Immuno-PET Using the Anti-CEA x Anti-HSG TF2 Bispecific Antibody and 68Ga-IMP-288 Peptide in Patients With Recurrences of Medullary Thyroid Carcinoma.
Brief Title: ImmunoTEP for Patients With Medullary Thyroid Carcinoma.
Acronym: iTEP-CMT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROG/10/94
Record Dates: First submitted 2012-11-12; First posted 2012-11-21 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2017-05

CONDITIONS: Medullary Thyroid Carcinoma
Keywords: thyroid,; endocrine tumour; Nuclear medicine,; molecular imaging; ImmunoTEP
MeSH Terms: conditions — Carcinoma, Medullary; Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TF2 antibody/68Ga-IMP-288 (Experimental): TF2 coupled with 68 Ga-IMP-288
  Interventions: Drug: • TF2 and 68 Ga-IMP-288

INTERVENTIONS:
Drug: • TF2 and 68 Ga-IMP-288
  Other Names: • TF2: trivalent recombinant humanized antibody recognizing the ACE and the peptide histamine-succinyl-glycine IMP-288 (HSG); • 68 Ga-IMP-288: di-HSG peptide-DOTA-labeled with Gallium 68

SUMMARY:
The aim of this study is to optimize pretargeting parameters using pharmacokinetic and imaging data for immuno-PET using anti-CEA x anti-HSG TF2 BsMAb and 150 MBq of 68Ga-IMP-288 peptide in MTC patients with abnormal Ct serum level after initial complete surgery and at least one abnormal lesion

DETAILED DESCRIPTION:
Variation of TF2 molar dose, IMP-288 molar dose and pretargeting interval will be performed in 4 to 5 cohorts of 3 patients, receiving 30 to 120 nmol of TF2 and 1.5 to 6 nmol of peptides 1 to 3 days apart. Blood samples will be obtained after TF2 and 68Ga-IMP-288 injections.

A last cohort (cohorte number 5 or 6) with optimal conditions will be proposed. Whole-body PET images will be recorded 60 and 120 minutes after 68Ga-IMP-288 injection to assess semi-quantitatively tumor targeting and tumor/background ratio. Moreover, the targeting sensitivity of the TF2-pretargeted 68Ga-IMP-288 will be compared to standard methods of tumor.

some patient will have a second immuno-TEP for their follow up in the first examen was the most sensible.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of CMT
* Calcitonin> 150 pg / ml
* Complete treatment of the primary tumor
* at least one detectable lesion more than 10 mm on conventional imaging: bone lesions can be taken into account if they extend outside of the bone and the party extra bone is measurable.
* Age ≥ 18 years
* Negative pregnancy test for women of childbearing age in the previous 2 days immuno-PET. Women of childbearing potential should use effective contraception take continuously for 3 months.
* KPS ≥ 70 or ECOG 0-1 and life expectancy of at least 6 months
* Absence of serious illness or co-morbidity assessed risk
* Creatinine ≤ 2.5 normal
* Absence of cancer treatment within 6 weeks prior to the immuno-PET
* No history of cancer within 5 years, except skin cancer other than melanoma or carcinoma in situ of the cervix
* Lack of anti-antibodies in patients who have previously received antibodies and hypersensitivity to antibody or protein
* Informed consent signed
* Social Insurance

Exclusion Criteria:

* Pregnancy or breastfeeding
* Serious illness or co-morbidity assessed risk
* History of cancer within 5 years, except skin cancer other than melanoma or carcinoma in situ of the cervix
* Presence of anti-antibodies in patients who have previously received antibodies
* Known hypersensitivity to antibody or protein
* Need to establish a cancer treatment within 3 months of immuno-PET (before stock evaluation 3 months)
* Inability intellectual sign consent
* Patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the tumor targeting (No Unit) and signal/noise (No Unit)ratio by immunoTEP with TF2 and 68-Ga-IMP-288 | one week
  Decrease of TF2 and IMP- 288 molar doses and variation of pretargeting interval will be performed in 4 to 5 cohorts of 3 patients, receiving 120 to 30 nmol of TF2 and 6 à 1.5 nmol of peptides 1 to 3 days apart.
  A last cohort (number 5 or 6) with optimal conditions will be proposed Blood samples will be obtained after TF2 and 68Ga-IMP-288 injections. Whole-body PET images will be recorded 60 to 120 minutes after 68Ga-IMP-288 injection to assess semiquantitatively tumor targeting and tumor/background ratio.

SECONDARY OUTCOMES:
Sensibilité | 6 monts after immunoTEP

OTHER OUTCOMES:
tolerance | 6 monts after immunoTEP
a second _iTEP if necessary for the follow up of a lesion | 6 monts after immunoTEP
  with in the follow up of the pateint

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Bodere, PhD, MD, Principal Investigator — Nantes Hospital
Locations (3):
- France (3):
  - Angers Hospital, Angers
  - Nantes Hospital, Nantes
  - Institut de Cancérologie de l'ouest, René Gauducheau, Saint-Herblain